CLINICAL TRIAL: NCT06738849
Title: EkiYou-Study-2 : Multicenter Randomised Controlled Trial of the EkiYou Application for Insulin Bolus Calculation
Brief Title: EkiYou-Study-2 : A National Multicentric Trial of the EkiYou Application for Insulin Bolus Calculation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: DiappyMed (Industry)
Collaborators: Sanoia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-A01531-46
Record Dates: First submitted 2024-12-04; First posted 2024-12-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Diabetes Type 1; Diabetes Type 2 on Insulin; Pancreatogenous Diabetes
Keywords: decision support system; digital therapy; bolus advisor; flexible insulin therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: the control group will switch to the interventional device after the first three months of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm (Experimental): The interventional device EkiYou V2 will be used at inclusion following randomization.
  Interventions: Device: EkiYou V2
- Control Arm (No Intervention): Control arm with standard care for the first three months. Participants use their standard basal bolus management method by fixed doses or flexible insulin therapy.
  After the initial three-months control period, participants will benefit from the investigational device EkiYou V2.

INTERVENTIONS:
Device: EkiYou V2 — Use of a Digital Therapy in the form of a mobile application that helps users to evaluate their daily bolus and basal insulin needs, and that adjusts at weekly basis their insulin to carb ratios, correction factor and basal dose.
  The device includes the following features to participants:
  * Carbohydrate counting through an extensive food database with more than 200k items.
  * Bolus calculation based on their meal, physical activity and blood glucose.
  * Bolus correction advice.
  * Long-acting insulin reminders and automatic periodic titration.
  * Insulin-to-carb ratios and correction factor automatic adjustment.
  Arms: Intervention Arm

SUMMARY:
EkiYou-Study-2 is an interventional multicenter randomised controlled clinical investigation according to EU 2017/745. It is conducted in 154 adults with diabetes and treated by multiple daily insulin injections that will be followed for 6 months.

After a randomization, participants will receive for 6 months EkiYou V2 Digital Therapy that will help them to estimate their daily bolus and basal insulin doses. This device weekly adjusts insulin parameters including : basal insulin dose, insulin to carb ratios and correction factor.

The control group will stay with their standard care, and after the first three months of control period, they will receive EkiYou V2 for the last three months.

The aim of this study is to examine the performance of the EkiYou V2 Digital Therapy compared with conventional methods for people with diabetes treated with multi-injections as part of a basal-bolus regimen. We also aim to assess the level of satisfaction and user experience with the EkiYou application, as well as the quality of life of study participants.

DETAILED DESCRIPTION:
Participants of the study must be adults treated with multiple daily insulin injections in a basal/bolus insulin regimen and users of a continuous glucose monitor (CGM). The study involves 3 visits (including the inclusion visit), for a total duration of 6 months for each participant.

The study participants will be randomized in two groups and will receive EkiYou V2 either at inclusion or at the second visit after three-months control period.

EkiYou V2 device is a new version of the previously CE-Marked device EkiYou V1. It is a decision support that include the following features to participants:

* Carbohydrate counting through an extensive food database with more than 200k items.
* Bolus calculation based on their meal, physical activity and blood glucose.
* Bolus correction advice.
* Long-acting insulin reminders and automatic periodic titration.
* Insulin-to-carb ratios and correction factor automatic adjustment.
* Connection to CGM devices

Participants will also respond to ePRO questionnaires during the clinical investigation to collect data on their quality of life and their satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* be aged 18 or over,
* have type 1 or type 2 diabetes or diabetes secondary to pancreatic disease,
* have been treated with multi-injection basal/bolus insulin therapy for at least 6 months,
* using a compatible rapid insulin with the device Ekiyou such as : Novorapid, Humalog, Apidra, Asparte Sanofi, Fiasp or Lyumjev,
* using a compatible long-acting insulin with the device EkiYou such as : Lantus, Abasaglar, Toujeo, Levemir or Tresiba,
* have been using a continuous glucose monitoring device such as Dexcom G6, Dexcom One, Dexcom One+ or FreeStyle Libre for at least 3 months,
* have given their physician access to their glucose data via a glucose data management platform,
* for type 2 diabetic patients using an hypoglycemia-inducing agent other than insulin (including hypoglycemic sulfonamides and SGLT-2 inhibitors), have no change in dosage regimen for at least 3 months
* have recorded at least 70% of CGM data over a 14-day window close to the inclusion date,
* have at least one smartphone running Android 5.0 or higher or iOS 12.0 or higher connected to the internet and able to receive CGM data available to them on the day of the inclusion,
* able to read or use a smartphone with no visual impairment needing specific typography,
* for patients of childbearing potential, a pregnancy test must have been carried out prior to inclusion, or an effective and adequate method of contraception must be used,
* be affiliated to a French social security scheme.

Exclusion Criteria:

* pregnant or breast-feeding women,
* type 1 diabetic patients treated with any hypoglycemia-inducing agent other than insulin (including hypoglycemic sulfonamides and SGLT-2 inhibitors),
* insulin-resistant patient: prescribed daily insulin dose > 1 U/kg/day or > 200 U/day,
* patient with very low insulin requirements: daily insulin dose < 15 U/day,
* patient with gastroparesis,
* diabetic ketoacidosis or severe level 3 hypoglycemia requiring third-party intervention within the 6 months prior to inclusion,
* pancreatic disease secondary to chronic ethanolism,
* known medical condition that, in the investigator's opinion, may interfere with the protocol,
* patient who cannot be monitored for 3 months,
* intellectual ability compromising use of the application, comprehension or completion of questionnaires,
* participation in another clinical trial or administration of a non-authorised drug in the 4 weeks preceding the screening,
* person taking part in another research study with an exclusion period still in progress,
* under guardianship or curatorship,
* imprisoned or otherwise deprived of liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in the percentage of time in range 70-180 mg/dL | At three Month Versus Inclusion
  Time in range is the amount of time spent in the target glucose range-between 70 and 180 mg/dL-as measured by CGM

SECONDARY OUTCOMES:
Number of non-serious adverse events related or unrelated to the device | Through study completion, an average of 6 months
  Severe hypoglycemia (Level 3) with blood glucose below 54 mg/dL and requiring assistance from an external person for carbohydrates intake or glucagon use.
Number of non-serious adverse events related or unrelated to the device | Through study completion, an average of 6 months
  Severe hyperglycemia (Level 3) defined by the presence of ketonemia > 3 mmol/L or ketonemia > 1 mmol/L and requiring consultation with a healthcare professional.
Number of serious clinical adverse events (SAEs) | Through study completion, an average of 6 months
  Number of severe level 3 hypoglycemic events requiring hospitalization
Number of serious clinical adverse events (SAEs) | Through study completion, an average of 6 months
  Number of episodes of diabetic ketoacidosis requiring hospitalization
Change in the percentage of time below 54 mg/dL | At Month 3 and Month 6
  Percentage of time with glucose below 54 mg/dL as measured by CGM
Change in the percentage of time below 70 mg/dL | At Month 3 and Month 6
  Percentage of time with glucose below 70 mg/dL as measured by CGM
Change in the percentage of time above 180 mg/dL | At Month 3 and Month 6
  Percentage of time with glucose above 180 mg/dL as measured by CGM
Change in the percentage of time above 250 mg/dL | At month 3 and Month 6
  Percentage of time with glucose above 250 mg/dL as measured by CGM
Change in the Glucose Management Indicator (GMI) | At month 3 and Month 6
  GMI as measured by CGM
Change in Mean blood glucose level | At month 3 and Month 6
  Mean sensor glucose as measured by CGM
Change in Coefficient of variation of blood glucose | At month 3 and Month 6
  Coefficient of variation of blood glucose as measured by CGM
Diabetes Treatment Satisfaction Questionnaire (DTSQ) | At month 3 and Month 6
  Quality of life associated with diabetes questionnaire
EQ-5D-5L questionnaire | At month 3 and Month 6
  Quality of life associated with diabetes questionnaire
ADDQoL-19 questionnaire | At month 3 and Month 6
  Quality of life associated with diabetes questionnaire

CONTACTS AND LOCATIONS:
Locations (16):
- France (16):
  - APHP Avicennes, Bobigny
  - CHU CAEN, Caen
  - IDNC, Chartres
  - CHSF Corbeil-Essonnes, Corbeil-Essonnes
  - Cabinet Dr Picard, Dijon
  - GH Le Havre - Hôpital Jacques Monod, Le Havre
  - CHU Limoges - Dupuytren, Limoges
  - Fondation Ambroise Paré / HEM, Marseille
  - Cabinet Dr Navaranne, Mérignac
  - University Hospital, Montpellier, Montpellier
  - APHP - Hôpital La Pitié Salpêtrière, Paris
  - CH Périgueux, Périgueux
  - Cabinet Dr Diedisheim, Saint-Cyr-sur-Loire
  - Cabinet Dr Gervaise, Saint-Cyr-sur-Loire
  - CHU Toulouse - Hôpital Rangueil, Toulouse
  - Clinique Pasteur, Toulouse

IPD SHARING:
Plan to Share IPD: No